CLINICAL TRIAL: NCT05361733
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, First-in-Human Study of the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of XFB19 in Healthy Adult Volunteers.
Brief Title: A First in Human Study of the Safety, Tolerability, and the Physiologically Based Pharmacokinetics of XFB19 in Healthy Adult Volunteers.
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Xfibra, Inc. (Industry)
Collaborators: PharPoint Research, Inc. (Industry); Safe Harbor Pharmacovigilance (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XFB19-101; HT94252510985 (Log # PR241349) (Other Grant/Funding Number: Department of Defense.)
Record Dates: First submitted 2022-04-08; First posted 2022-05-05 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Focus of the Study: Safety of XFB19
Keywords: human C/EBPβ-Thr266; XFB19

STUDY DESIGN:
Intervention Model Description: In Part A, 24 healthy volunteers will be enrolled in a total of 3 cohorts (Cohorts A1 to A3) with ascending doses of XFB19: 5mg (Cohort A1), 10mg (Cohort A2), and 20mg (Cohort A3). Each cohort will enroll 8 participants with 6 participants randomized to receive XFB19 and 2 participants randomized to receive placebo.
  In Part B, 16 healthy volunteers will be enrolled in a total of 2 cohorts (Cohorts B1 and B2). Each cohort will enroll 8 participants with 6 participants randomized to receive XFB19 and 2 participants randomized to receive placebo. Cohorts B1 and B2 will accept the second highest and highest XFB19 doses for evaluation from Part A.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Sponsor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- XFB19 administered SC. (Experimental): Part A: XFB19 SC injection at the following dose levels:
  * Cohort A1: 5 mg (or placebo vehicle , same volume)
  * Cohort A2: 10 mg (or placebo vehicle , same volume)
  * Cohort A3: 20 mg (or placebo vehicle , same volume)
  Part B: XFB19 SC injection at the 2 highest acceptable dose levels from Part A:
  * Cohort B1: second highest acceptable dose level from Part A (or placebo vehicle , same volume)
  * Cohort B2: highest acceptable dose level from Part A (or placebo vehicle , same volume)
  Interventions: Drug: XFB19
- Placebo (Placebo Comparator): 10 healthy volunteers will be randomized and assigned to the Placebo arm in Part A (Cohorts A1, A2 and A3) and Part B (Cohorts B1 and B2).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XFB19 — The site-specific phosphorylation of the CCAAT/enhancer binding protein β (C/EBPβ) on Threonine266 (phospho-C/EBPβThr266) is critical for the priming and activation pathways, signals 1 and 2 of the NLRP3 inflammasome, that result in its full induction, causal to systemic inflammation critical to the morbidity and mortality of inflammatory/fibrotic diseases.
  Phospho-C/EBPβThr266 is also essential for the mesenchymal myofibroblastic cell cycle checkpoint failure and transition that results in the inappropriate tissue repair and pathological tissue fibrosis.
  XFB19 is a first-in-class, rationally-designed drug. It is homeostatic, and in preclinical studies, effectively, safely, and selectively inhibits phospho-C/EBPβThr266, the pathological inflammatory-fibrotic complications of NLRP3 inflammasome activation and synergistic myofibroblastic transition, reversing the pathology towards homeostasis, and fulfilling the precision medicine objectives.
  Arms: XFB19 administered SC.
Drug: Placebo — No active ingredient drug use to blind participants and investigators
  Arms: Placebo

SUMMARY:
Xfibra, Inc. is conducting a Phase 1, randomized, double-blind, placebo-controlled, first-in-human study of the safety, tolerability, and physiologically-based pharmacokinetics (PK) of single and multiple ascending doses of XFB19 in healthy adult volunteers.

DETAILED DESCRIPTION:
Xfibra, Inc. is conducting this clinical research study to test a potential new drug called XFB19 that is being developed for inflammatory/fibrotic diseases.

Although current medications are available to improve health and survival in patients with inflammatory/fibrotic diseases no specific pharmacotherapy has proven curative against Acute Respiratory Distress Syndrome (ARDS), liver cirrhosis , or Idiopathic Pulmonary Fibrosis (IPF). The advantages of XFB19 over currently available therapies are its target specificity, in that it only affects a carefully selected target which may allow recovery from inflammatory/fibrotic diseases, and potentially reverse tissue fibrosis.

Although many laboratory and animal studies have been completed, this is the first time XFB-19 is being tested in humans. Therefore, side effects in humans are unknown.

This study will be conducted in two parts - Part A (single dose) and Part B (multiple dosing). The purpose and main goals of this study are:

* To determine whether XFB19 is safe and well tolerated in humans
* To determine a safe dose of XFB19 to be used in future studies in patients.
* To test how much XFB19 gets into the blood and how long it takes to be cleared from the body
* To measure the activity of XFB19 in blood.

XFB19 is considered experimental because it has not yet been approved by the FDA (Food and Drug Administration) in the USA, or any other regulatory agency responsible for approving medicines. There may be risks in taking this experimental drug that are unknown.

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the study, including possible risks and adverse effects.
2. Adult males and females, 18 to 55 years of age (inclusive) at screening.
3. Body mass index ≥ 18.0 and ≤ 35.0 kg/m2 with a body weight ≥ 45 kg at screening.
4. Be non-smokers (including tobacco, e-cigarettes, and marijuana) for at least 1 month prior to first investigational drug administration.
5. Medically healthy without clinically significant abnormalities (in the opinion of the Investigator) at the Screening Visit and prior to dosing including:

   1. Physical examination without any clinically significant findings
   2. Systolic blood pressure in the range of 90 to 160 mmHg (inclusive) and diastolic blood pressure in the range of 50 to 95 mmHg (inclusive) after 5 minutes rest in supine position
   3. Heart rate (HR) in the range of 40 to 100 bpm (inclusive) after 5 minutes rest in supine position
   4. Body temperature (tympanic or oral) in the range of 35.5°C to 37.7°C (inclusive)
   5. No clinically significant findings in serum chemistry, hematology, coagulation, and urinalysis tests
   6. Triplicate 12-lead ECGs (taken after the volunteer has been supine for at least 5 minutes) with QT intervals corrected using Fridericia's method (QTcF) ≤ 450 msec for males and ≤ 470 msec for females and no clinically significant abnormalities
6. Female volunteers must:

   1. Be of nonchildbearing potential, i.e., surgically sterilised (hysterectomy, bilateral salpingectomy, bilateral tubal ligation, bilateral oophorectomy at least 6 weeks before screening) or postmenopausal (defined as no menses for 12 months without an alternative medical cause and a follicle-stimulating hormone [FSH] level > 40 IU/L at the Screening Visit) OR
   2. If of childbearing potential, must agree not to donate ova, not to attempt to become pregnant, and, if engaging in sexual intercourse with a male partner, must agree to use an acceptable method of contraception from the time of signing the participant informed consent form (PICF) until at least 30 days after the last dose of the study drug
7. Male volunteers must agree not to donate sperm, and, if engaging in sexual intercourse with a female partner who could become pregnant, must agree to use an acceptable method of contraception from the time of signing the consent form until at least 30 days after the last dose of study drug.
8. Have suitable venous access for blood sampling.
9. Be willing and able to comply with all study assessments and adhere to the protocol schedule and restrictions.

Exclusion Criteria:

1. History or presence of any clinically significant (as determined by the PI) cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, or neurological disease, including any acute illness or major surgery, within the past 3 months.
2. Current infection that requires systemically absorbed antibiotic, antifungal, antiparasitic, or antiviral medications.
3. Any history of malignant disease in the last 5 years (excluding surgically resected skin squamous cell or basal cell carcinoma).
4. Presence of clinically relevant immunosuppression from, but not limited to, immunodeficiency conditions such as common variable hypogammaglobulinemia.
5. Use of or plans to use systemic immunosuppressive (e.g., corticosteroids, methotrexate, azathioprine, cyclosporine) or immunomodulating medications (e.g., interferon) during the study or within 3 months prior to the first study drug administration.
6. History of risk factors for torsade de pointes (including a family history of long QT syndrome or sudden cardiac death) or a known arrythmia.
7. Liver function test (LFT) results > 1.5 times the upper limit of normal (ULN) for gamma glutamyl transferase (GGT), bilirubin (total, conjugated, and unconjugated), alkaline phosphatase (ALP), aspartate aminotransferase (AST), or alanine aminotransferase (ALT). Volunteers with bilirubin, ALP and/or ALT/AST above the limits specified may be included, at the discretion of the Investigator, if the levels are unaccompanied by clinical signs.
8. Positive test results for human immunodeficiency virus (HIV-1 or HIV-2) antibodies, hepatitis C virus (HCV) antibodies, or hepatitis B surface antigen (HBsAg) at the Screening Visit. Patients with HCV antibodies, or HBsAg could be included if the viral load for HCV or hepatitis B are negative.
9. Positive test result for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) via polymerase chain reaction or commercially validated antigen test, per site's standard clinical procedure.
10. Presence of sequelae of gastrointestinal, liver, kidney, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
11. Estimated creatinine clearance (CrCl) < 60 mL/min using the Cockcroft-Gault formula or serum creatinine more than 1.5 x ULN.
12. History of substance abuse or alcohol abuse (defined as more than 10 standard drinks per week or regularly consuming more than 4 standard drinks per day where 1 standard drink is 10 g of pure alcohol and equivalent to 285 mL beer [4.9% Alc./Vol], 100 mL wine [12% Alc./Vol], or 30 mL spirit [40% Alc./Vol]) within 12 months prior to the Screening Visit.
13. Positive drugs of abuse or alcohol breath test results at the Screening Visit or at CRU check in (Day -1) (repeat tests allowed if false positive suspected). Non-habitual use and agreement to refrain from using any THC/CBD products during the study is allowed.
14. Use of any prescription or over the counter (OTC) medication (including herbal products, diet aids, and hormone supplements) within 10 days or 5 half-lives of the medication (whichever is longer) prior to the first study drug administration, excepting use of contraceptives and occasional use of acetaminophen (up to 1 g every 8 hours or 3 g per day maximum).
15. Demonstrated clinically significant (required intervention, e.g., emergency room visit, epinephrine administration) allergic reactions (e.g., food, drug, or atopic reactions, asthmatic episodes) which, in the opinion of the Investigator, would interfere with the volunteer's ability to participate in the study.
16. Known hypersensitivity to any of the study drug ingredients.
17. Use of any vaccinations within 10 days prior to first study drug administration.
18. For women of childbearing potential, a positive serum pregnancy test at the Screening Visit or a positive urine pregnancy test (with confirmatory positive serum pregnancy test) at CRU check-in (Day -1).
19. Currently breastfeeding.
20. Donation of blood or plasma or loss of whole blood of more than 500 mL within 30 days prior to first study drug administration or receipt of a blood transfusion within 2 months prior to first study drug administration.
21. Participation in another clinical study of an investigational drug within 30 days or 5 half-lives of the investigational agent (whichever is longer) prior to the first study drug administration.
22. Any other condition or prior therapy that in the opinion of the Investigator would make the volunteer unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol or likelihood of noncompliance with any study requirements.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | During admission to the clinical unit (up to 10 days)
  Number of participants with adverse events (using the CTCAE v5.0 grading scale), with abnormal laboratory tests results (hematology, serum chemistry, coagulation, and urinalysis), abnormal vital signs, abnormal ECG parameters, and abnormal physical examination findings.
Heart Rate (assessed by ECG) | During admission to the clinical unit (up to 10 days)
  ECG parameters include the following:
  Heart Rate
Rhythm (assessed by ECG) | During admission to the clinical unit (up to 10 days)
  ECG parameters include the following:
  Rhythm
P wave (assessed by ECG) | During admission to the clinical unit (up to 10 days)
  ECG parameters include the following:
  P wave
PR interval (assessed by ECG) | During admission to the clinical unit (up to 10 days)
  ECG parameters include the following:
  PR interval
QRS complex (assessed by ECG) | During admission to the clinical unit (up to 10 days)
  ECG parameters include the following:
  QRS complex
ST segment (assessed by ECG) | During admission to the clinical unit (up to 10 days)
  ECG parameters include the following:
  ST segment
T wave (assessed by ECG) | During admission to the clinical unit (up to 10 days)
  ECG parameters include the following:
  T wave
QT interval (assessed by ECG) | During admission to the clinical unit (up to 10 days)
  ECG parameters include the following:
  QT interval
Cardiac axis (assessed by ECG) | During admission to the clinical unit (up to 10 days)
  ECG parameters include the following:
  Cardiac axis
J-point (assessed by ECG) | During admission to the clinical unit (up to 10 days)
  ECG parameters include the following:
  J-point

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) | During admission to the clinical unit (up to 10 days)
  XFB19 PK endpoints include (but are not limited to) the following after the single dose in Part A and/or the first and last doses in Part B as indicated:
  • Cmax
Time to Cmax (Tmax) | During admission to the clinical unit (up to 10 days)
  XFB19 PK endpoints include (but are not limited to) the following after the single dose in Part A and/or the first and last doses in Part B as indicated:
  • Tmax
Trough concentration (Ctrough) | During admission to the clinical unit (up to 10 days)
  XFB19 PK endpoints include (but are not limited to) the following after the single dose in Part A and/or the first and last doses in Part B as indicated:
  • Ctrough (predose Day 7 in Part B only)
Area under the plasma drug concentration-time curve (AUC0-tlast). | During admission to the clinical unit (up to 10 days)
  XFB19 PK endpoints include (but are not limited to) the following after the single dose in Part A and/or the first and last doses in Part B as indicated:
  • Area under the plasma drug concentration-time curve from time zero to the time of last quantifiable concentration (AUC0-tlast)
Apparent terminal elimination half-life (t1/2) | During admission to the clinical unit (up to 10 days)
  XFB19 PK endpoints include (but are not limited to) the following after the single dose in Part A and/or the first and last doses in Part B as indicated:
  • t1/2
Apparent terminal elimination half-life (t1/2) | During admission to the clinical unit (up to 10 days)
  XFB19 PK endpoints include (but are not limited to) the following after the single dose in Part A and/or the first and last doses in Part B as indicated:
  • Apparent terminal elimination half-life (t1/2)
Terminal elimination rate constant (λz) | During admission to the clinical unit (up to 10 days)
  XFB19 PK endpoints include (but are not limited to) the following after the single dose in Part A and/or the first and last doses in Part B as indicated:
  • λz
Total apparent body clearance (CL/F) | During admission to the clinical unit (up to 10 days)
  XFB19 PK endpoints include (but are not limited to) the following after the single dose in Part A and/or the first and last doses in Part B as indicated:
  • CL/F
Apparent volume of distribution (Vz/F) | During admission to the clinical unit (up to 10 days)
  XFB19 PK endpoints include (but are not limited to) the following after the single dose in Part A and/or the first and last doses in Part B as indicated:
  • Vz/F
Apparent steady state volume of distribution (Vss/F) | During admission to the clinical unit (up to 10 days)
  XFB19 PK endpoints include (but are not limited to) the following after the single dose in Part A and/or the first and last doses in Part B as indicated:
  • Vss/F

OTHER OUTCOMES:
Transcriptome in blood cells. | During admission to the clinical unit (up to 10 days)
  Transcriptome in blood cells will be analyzed by RNA sequencing . The results of these analyses will be summarized by treatment.
Inflammatory proteins in blood. | During admission to the clinical unit (up to 10 days)
  Inflammatory protein in blood will be analyzed by cytokine/chemokine multiplex assay. The results of these analyses will be summarized by treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Martina M Buck, Ph.D., Study Chair — Xfibra, Inc.

IPD SHARING:
Plan to Share IPD: No
No at this time, as Xfibra, Inc. will evaluate data internally and may share data at a later time period.

REFERENCES:
- [Background] Buck M, Chojkier M. A ribosomal S-6 kinase-mediated signal to C/EBP-beta is critical for the development of liver fibrosis. PLoS One. 2007 Dec 26;2(12):e1372. doi: 10.1371/journal.pone.0001372. PMID 18159255
- [Background] Buck M, Chojkier M. C/EBPbeta associates with caspase 8 complex proteins and modulates apoptosis in hepatic stellate cells. J Clin Gastroenterol. 2007 Nov-Dec;41 Suppl 3:S295-9. doi: 10.1097/MCG.0b013e31814927d5. PMID 17975479
- [Background] Buck M, Chojkier M. C/EBPbeta-Thr217 phosphorylation signaling contributes to the development of lung injury and fibrosis in mice. PLoS One. 2011;6(10):e25497. doi: 10.1371/journal.pone.0025497. Epub 2011 Oct 5. PMID 21998664
- [Background] Buck M, Poli V, Hunter T, Chojkier M. C/EBPbeta phosphorylation by RSK creates a functional XEXD caspase inhibitory box critical for cell survival. Mol Cell. 2001 Oct;8(4):807-16. doi: 10.1016/s1097-2765(01)00374-4. PMID 11684016
- [Background] Buck M, Solis-Herruzo J, Chojkier M. C/EBPbeta-Thr217 Phosphorylation Stimulates Macrophage Inflammasome Activation and Liver Injury. Sci Rep. 2016 Apr 12;6:24268. doi: 10.1038/srep24268. PMID 27067260